CLINICAL TRIAL: NCT06245746
Title: A Single-center, Prospective Trial of the Safety and Efficacy of UCMSC-Exo in Consolidation Chemotherapy-induced Myelosuppression in Patients With Acute Myeloid Leukemia After Achieving Complete Remission
Brief Title: UCMSC-Exo for Chemotherapy-induced Myelosuppression in Acute Myeloid Leukemia
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Qiubai Li, M.D. & Ph.D., Professor, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UHCT231013
Record Dates: First submitted 2024-01-30; First posted 2024-02-07 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Acute Myeloid Leukemia; Neutropenia; Anemia; Thrombocytopenia; Infections; Bleeding
Keywords: umbilical cord derived mesenchymal stem cells exosomes; chemotherapy-induced myelosuppression; neutropenia; anemia; thrombocytopenia; infections; bleeding; acute myeloid leukemia; chemotherapy
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Neutropenia; Anemia; Thrombocytopenia; Infections; Hemorrhage

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- UCMSC-Exo intervention (Experimental): UCMSC-Exo will be preset with 3 escalation dose levels in single time infusion.
  Interventions: Biological: umbilical cord derived mesenchymal stem cells exosomes (UCMSC-Exo)

INTERVENTIONS:
Biological: umbilical cord derived mesenchymal stem cells exosomes (UCMSC-Exo) — UCMSC-Exo will be infused intravenously.

SUMMARY:
The purpose of the study is to explore the safety and efficacy of UCMSC-Exo in consolidation chemotherapy-induced myelosuppression in patients with acute myeloid leukemia after achieving complete remission.

DETAILED DESCRIPTION:
Despite the improved prognosis of patients with acute myeloid leukemia, almost all patients will experience severe myelosuppression induced by chemotherapy, leading to a series of complications such as infection due to neutropenia, bleeding due to thrombocytopenia and/or impaired major organ function such as cardiac function due to anemia, which are the main reasons for dose reduction, dose interruptions of chemotherapy and also treatment-related death. It is of significant clinical importance and an urgent need to promote early recovery of myelosuppression and reduce risks of related complications as well as medical burdens. Umbilical cord derived mesenchymal stem cells exosomes (UCMSC-Exo), as the key effector of the stem cells with multipotential, can widely act on the functional cell units of bone marrow microenvironment and promote the repairment and regeneration of key cells such as hematopoietic stem cells, mesenchymal stem cells and endothelial cells, thus making it an ideal means for effectively promoting recovery of myelosuppression. Patients with acute myeloid leukemia who have achieved complete remission (CR) and are going to receive consolidation chemotherapy will be invited to participate in the study, to receive UCMSC-Exo intravenous infusion and follow-up visits of up to 1 years after enrollment.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 18 and 60 years old;
2. Acute myeloid leukemia (AML, AML subtype M3 excluded) diagnosed according to the 2022 revision to the World Health Organization classification of myeloid neoplasms and acute leukemia, who have achieved complete remission (CR1) and are going to receive consolidation therapy (cytarabine or cytarabine-based combined regimen, the cycle of consolidation therapy is not limited);
3. The participant or his/her legal guardian is adequately informed of the nature and risks of the study, voluntarily participates in the study with signed informed consent;
4. Male or female;
5. Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 to 2 (by the day chemotherapy is initiated)
6. Estimated survival of at least 3 months;
7. Adequate major organ function:

   1. Respiratory function: indoor oxygen saturation of at least 95%;
   2. Cardiac function: ejection fraction of left ventricular of at least 45%;
   3. Hepatic function: alanine aminotransferase/aspartate aminotransferase of at most 2.5 times/upper limit of normal value and serum total bilirubin of at most 1.5 times/upper limit of normal value;
   4. Renal function: Serum creatinine of at most 1.5 times/upper limit of normal value;
8. Participants who do not receive any type of anti-cancer therapy within 2 weeks before enrollment (radiation therapy, chemotherapy and/or immune therapy, et al.), and treatment-associated toxicities induced by previous therapy has recovered to Grade 1 or below (except for low grade toxicities such as alopecia).
9. For female participants, they should be surgical sterilized or post-menopausal, or agree to utilize a medically recognised method of contraception (such as intrauterine device, condom) during treatment period of the study and within 6 months after the end of treatment period of the study; For male participants, they should be surgical sterilized or agree to utilize a medically recognised method of contraception (such as intrauterine device, condom) during treatment period of the study and within 6 months after the end of treatment period of the study;

Exclusion Criteria:

1. Central nervous system manifestations of acute myeloid leukemia at diagnosis;
2. Secondary acute myeloid leukemia;
3. Myelosuppression induced by conditions other than anti-cancer therapy;
4. Previous radiation therapy performed on sternum or pelvis;
5. Specifically diagnosed and uncontrolled infection at enrollment (Uncontrolled is defined as exhibiting ongoing signs and symptoms of infection without improvement despite anti-infective agents) ;
6. Uncontrolled active bleeding at enrollment;
7. Severe underlying comorbidities affecting survival, including cachexia, severe malnutrition, etc;
8. Estimated survival of at most 48 hours;
9. Active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection;
10. History of or current human immunodeficiency virus (HIV) infection;
11. Syphilis infection;
12. Continuous usage of immunosuppressants or received organ transplantation in the last 6 months;
13. Participation in clinical trials of other drugs within 6 weeks before enrollment;
14. Previous participation in clinical stem cell or exosome research;
15. Receive any agent concurrently with UCMSC-Exo infusion which inhibits cell division (hydroxyurea, low-dose cytarabine or methotrexate, etc) ;
16. Severe allergic constitution, or known or suspected allergy to the study drug and its components;
17. Known contraindication to receiving hematopoietic growth factors, transfusion of blood components, anti-infective agents;
18. Female participants who are pregnant or breast feeding;
19. Participants suffering from mental illness;
20. Presence of drug abuse/addiction;
21. History of other malignancies other than hematological malignancies within 3 years;
22. Participants without signed informed consent;
23. Participants with poor compliance and are unable to complete the whole course of the study;
24. Participants with circumstances that, in the opinion of the investigator, may increase the risk of the participants or interfere with conduct of the clinical trial and the judgment of results (excessive tension, sensitivity or cognitive impairment, etc) ;
25. Participants with other circumstances that are ineligible for enrollment in this study, in the opinion of the investigator.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9 (Estimated)
Dates: Start 2025-02-26 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events (AEs) and Serious Adverse Events (SAEs) | From the day that UCMSC-Exo is infused to up to 28 days (short-term safety follow-up) and 1 year (long-term safety follow-up)
  To investigate the safety characteristics, percentages will be calculated and grade will be evaluated.
Dose-limiting toxicities（DLT) | From the day that UCMSC-Exo is infused to up to 14 days
  During the DLT observation period, the subject has an adverse event that is reasonably related to UCMSC-Exo infusion (possibly, likely or definitely related).
Maximum tolerated dose (MTD) | From the day that UCMSC-Exo is infused to up to 14 days
  During the dose-escalation, the highest dose of dose-limiting toxicity for subjects no more than 1/6 in the dose group of at least 6 evaluable subjects of the study drug.

SECONDARY OUTCOMES:
Time to absolute neutrophil count recovery | From the start of chemotherapy to up to 42 days
  To investigate the efficacy characteristics, time will be measured in days.
Incidence of febrile neutropenia | From the start of chemotherapy to up to 42 days
  To investigate the efficacy characteristics, percentages will be calculated.
Duration of febrile neutropenia | From the start of chemotherapy to up to 42 days
  To investigate the efficacy characteristics, the duration will be measured in days.
Incidence of severe thrombocytopenia | From the start of chemotherapy to up to 42 days
  To investigate the efficacy characteristics, percentages will be calculated.
Time to severe thrombocytopenia recovery | From the start of chemotherapy to up to 42 days
  To investigate the efficacy characteristics, time will be measured in days.
Incidence of severe anemia | From the start of chemotherapy to up to 42 days
  To investigate the efficacy characteristics, percentages will be calculated.
Time to severe anemia recovery | From the start of chemotherapy to up to 42 days
  To investigate the efficacy characteristics, time will be measured in days.
Incidence of infection | From the start of chemotherapy to up to 42 days
  To investigate the efficacy characteristics, percentages will be calculated.
Duration of infection | From the start of chemotherapy to up to 42 days
  To investigate the efficacy characteristics, the duration will be measured in days.
Incidence of bleeding | From the start of chemotherapy to up to 42 days
  To investigate the efficacy characteristics, percentages will be calculated.
Duration of bleeding | From the start of chemotherapy to up to 42 days
  To investigate the efficacy characteristics, the duration will be measured in days.
Application rate of blood transfusion | From the start of chemotherapy to up to 42 days
  To investigate the efficacy characteristics, percentages will be calculated.
Application rate of anti-infective agents | From the start of chemotherapy to up to 42 days
  To investigate the efficacy characteristics, percentages will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Qiubai Li, Professor, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Wuhan Union Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No